CLINICAL TRIAL: NCT02077179
Title: Health Improvement After Pregnancy (HIP) Program Randomized Control Trial
Acronym: HIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor retention and recruitment,changes need to be made to the program
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Graeme Smith, Professor and Head of Obstetrics and Gynecology, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OBGY-249-14
Record Dates: First submitted 2014-02-26; First posted 2014-03-04 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Metabolic Cardiovascular Syndrome
Keywords: Postpartum; Preeclampsia; Gestational Hypertension; Gestational Diabetes; Exercise Intervention; Dietary Intervention; Behavioral Intervention; Mobile Website; Mobile Application
MeSH Terms: conditions — Metabolic Syndrome; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Participants in this arm will receive care as per the usual standards from Kingston General Hospital and their primary care provider.
- HIP Program (Experimental): Participants in this arm will follow the HIP Program in addition to their usual care from Kingston General Hospital and their primary care provider.
  Interventions: Behavioral: HIP Program

INTERVENTIONS:
Behavioral: HIP Program — The entirety of the HIP Program is delivered through an interactive mobile website.
  The physical activity portion of the program consists of daily step counting, prescribed aerobic activity, structured strength and toning workouts, and daily stretching. The program was designed by a local trainer, specializing in postnatal exercise, to increase gradually in intensity, while encouraging a more active lifestyle. The program is designed to be completed at home with minimal equipment.
  The nutrition portion of the program consists of 16 video tutorials developed by a local Registered Dietitian and weekly diet logs. The video tutorials cover all aspects of healthy eating, from the basics of Canada's Food Guide, to smart snacking, to eating healthy over the holidays.
  Arms: HIP Program

SUMMARY:
Recent Canadian studies, public opinion polls and the Canadian Heart Health Strategy and Action Plan state that women's heart health is a key national priority; it should be addressed through improving heart health awareness and prevention, and reducing care inequities for women in general and younger women in particular. The investigators have developed an innovative and interactive mobile website based postpartum lifestyle modification program (regular physical activity and nutritional guidance), based on established national guidelines, to improve heart disease risk factors in women. The investigators will conduct a trial to determine if the mobile website based lifestyle modification program can be maintained and reduces a collection of risk factors, which occurring together, greatly increases the risk of developing heart disease. The investigators hypothesize that the interactive mobile website directing regular physical activity and personalized nutritional guidance, compared to standard postpartum care, will be motivational and result in a reduced modified metabolic syndrome z score at 8 months postpartum among the intervention group.

ELIGIBILITY:
Inclusion Criteria:

- must own or have daily access to one or more of the following; smart phone, tablet or laptop computer

Exclusion Criteria:

* Living greater than 100km from Kingston General Hospital
* Having an existing and long term contraindication to exercise at the time of recruitment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Metabolic Syndrome Z Score | 32 weeks postpartum
  The primary outcome measure is the metabolic syndrome (MetS) z score, a continuous score of the five metabolic syndrome variables that make up the Adult Treatment Panel (ATP) III diagnostic criteria (waist circumference, blood pressure, high density lipoprotein, triglycerides and glucose). Differences between study arms will be compared.

SECONDARY OUTCOMES:
Adherence to the HIP Program; Percent of Workouts Completed | 32 weeks postpartum
  Adherence to the HIP Program will be assessed based on the number of times a participant indicates using the mobile website that a prescribed workout has been completed. This outcome will only be measured in the intervention arm.
Differences in Biochemical Cardiovascular Risk Markers | 32 weeks postpartum
  Differences between study arms for the following biochemical cardiovascular risk markers will be assessed at 32 weeks postpartum; lipid profile, fasting glucose, glycated hemoglobin, high sensitivity C-reactive protein, and urine microalbumin creatinine ratio.
Change in Anthropomorphic Measurements and Blood Pressure from Baseline at Midpoint | 20 weeks postpartum
  Changes in systolic blood pressure, diastolic blood pressure and weight from baseline measures at 6-8 weeks postpartum will be assessed at the midpoint of the program at 20 weeks postpartum. Differences between study arms will be compared.
Change in Anthropomorphic Measurements and Blood Pressure from Baseline at Study Completion | 32 weeks postpartum
  Changes in systolic blood pressure, diastolic blood pressure and weight from baseline measures at 6-8 weeks postpartum will be assessed at the midpoint of the program at 32 weeks postpartum. Differences between study arms will be compared.
Change in Anthropomorphic Measurements and Blood Pressure from Midpoint to Study Completion | 32 weeks postpartum
  Changes in systolic blood pressure, diastolic blood pressure, weight, body mass index, hip circumference, and waist circumference from midpoint measures at 20 weeks postpartum will be assessed at the end of the program at 32 weeks postpartum. Differences between study arms will be compared.
Adherence to the HIP Program; Percent of Step Counting Completed | 32 weeks postpartum
  Adherence to the HIP Program will be assessed based on the number of times a participant uses the mobile website to log their daily step count total. The number of times that the logged step count meets or exceeds the prescribed number of daily steps will also be assessed. This outcome will only be measured in the intervention arm.
Adherence to the HIP Program; Percent of Dietary Logs Completed | 32 weeks postpartum
  Adherence to the HIP Program will be assessed based on the number of times a participant uses the mobile website to enter the weekly dietary log. The number of times that the dietary log meets the prescribed intake for each of the Canada's Food Guide food groups will also be assessed. This outcome will only be measured in the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme N Smith, MD,PhD,FRCSC, Principal Investigator — Queen's University
Locations (1):
- Queen's Unviersity, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith GN, Pudwell J, Roddy M. The Maternal Health Clinic: a new window of opportunity for early heart disease risk screening and intervention for women with pregnancy complications. J Obstet Gynaecol Can. 2013 Sep;35(9):831-839. doi: 10.1016/S1701-2163(15)30841-0. No abstract available. PMID 24099450
- [Background] Cusimano MC, Pudwell J, Roddy M, Cho CK, Smith GN. The maternal health clinic: an initiative for cardiovascular risk identification in women with pregnancy-related complications. Am J Obstet Gynecol. 2014 May;210(5):438.e1-9. doi: 10.1016/j.ajog.2013.12.001. Epub 2013 Dec 4. PMID 24316270
- [Background] Smith GN, Pudwell J, Walker M, Wen SW. Risk estimation of metabolic syndrome at one and three years after a pregnancy complicated by preeclampsia. J Obstet Gynaecol Can. 2012 Sep;34(9):836-841. doi: 10.1016/S1701-2163(16)35382-8. PMID 22971452
- [Background] Smith GN, Pudwell J, Walker M, Wen SW. Ten-year, thirty-year, and lifetime cardiovascular disease risk estimates following a pregnancy complicated by preeclampsia. J Obstet Gynaecol Can. 2012 Sep;34(9):830-835. doi: 10.1016/S1701-2163(16)35381-6. PMID 22971451
- [Background] Smith GN, Walker MC, Liu A, Wen SW, Swansburg M, Ramshaw H, White RR, Roddy M, Hladunewich M; Pre-Eclampsia New Emerging Team (PE-NET). A history of preeclampsia identifies women who have underlying cardiovascular risk factors. Am J Obstet Gynecol. 2009 Jan;200(1):58.e1-8. doi: 10.1016/j.ajog.2008.06.035. Epub 2008 Aug 8. PMID 18691690